CLINICAL TRIAL: NCT01071616
Title: Oral Fluid, Plasma and Whole Pharmacokinetics and Stability Following Smoked Cannabis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 999910458; 10-DA-N458
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2013-11-29

CONDITIONS: Cannabis Use; Drug Abuse
Keywords: Cannabinoids; Oral Fluid; Pharmacokinetics; Stability; Smoked Cannabis
MeSH Terms: conditions — Substance-Related Disorders

INTERVENTIONS:
Drug: Cannabis Cigarette

SUMMARY:
Background:

- Little research has been done on how different components of cannabis (marijuana) appear in oral fluid (i.e., saliva) after smoking. Cannabinoids have been well studied in whole blood, plasma, and urine after cannabis use, but less is known about how cannabinoids appear in oral fluid after controlled drug administration and how long these biomarkers last after use. In addition, the issue of stability of cannabinoids and their glucuronide metabolites is a controversial topic that is poorly understood. These data are critical to the interpretation of cannabinoid test results.

Objectives:

* To collect whole blood, plasma, urine, and oral fluid specimens after smoking cannabis, to characterize the disposition and pharmacokinetics of cannabinoids in multiple biological matrices and to provide scientifically reliable data on the stability of cannabinoids and metabolites.
* To test basic brain function and thinking processes after smoking cannabis.

Eligibility:

- Healthy volunteers between 18 and 45 years of age who use cannabis (an average of at least twice per month in the 3 months before the study.)

Design:

* Participants may complete the single study session as outpatients, or they may spend the night prior to and/or following drug administration at the residential research unit in Baltimore, MD. Participants must provide a negative urine drug screen if they have not spent the evening prior to testing at the research unit.
* Participants will provide whole blood, plasma, oral fluid, and urine samples, and will complete several tests of thinking and brain function at the start of the study.
* Participants will smoke one standardized cannabis cigarette. Blood and oral fluid samples will be collected, and participants will repeat the tests of thinking and brain function multiple times after smoking.
* Six hours after smoking the cigarette, participants must pass a neuromotor exam (testing balance and coordination) before they can be discharged from the study. Participants may be asked to stay overnight at the clinical center if there are concerns for their safety because of intoxication.

DETAILED DESCRIPTION:
Background: Smoking is the most common route of cannabis administration, yet the pharmacokinetic properties of cannabinoids in oral fluid following cannabis smoking have not been adequately characterized. Characterization of cannabinoid pharmacokinetics in oral fluid, correlations between concentrations in different matrices and relationships between biomarker concentrations and concurrent pharmacodynamic effects are critical for the appropriate interpretation of cannabinoid tests. Furthermore, the short- and long-term stability of cannabinoid biomarkers, including glucuronide conjugates, in authentic whole blood, plasma, and oral fluid specimens following cannabis smoking is poorly defined. The only stability data available are from fortified samples, rather than authentic specimens.

Objectives: Part A: (1) Characterize cannabinoid ( -9-tetrahydrocannabinol, [THC]; 11-hydroxy-THC, [11-OH-THC]; 11-nor-9-carboxy-THC, [THCCOOH]; and their Phase II conjugates) pharmacokinetics in whole blood, plasma, oral fluid and urine following a single smoked dose of cannabis. (2) Determine inter-matrix cannabinoid ratios in authentic specimens following controlled smoked cannabis (3) Correlate cannabinoid concentrations in whole blood, plasma and oral fluid with impairment and risk-taking behavior as determined through subjective assessments, risk-behavior trait assessments and neurocognitive tasks. (4) Determine stability over time of free and conjugated cannabinoids in authentic whole blood, plasma, and oral fluid from cannabis users following a single smoked dose of cannabis under various storage conditions. (5) Characterize the sensitivity, specificity, efficiency and duration of detection of cannabinoids with the Draeger DrugTest 5000 after a single smoked dose of cannabis.

Part B: Characterize cannabinoid pharmacokinetics in whole blood, plasma, oral fluid, breath, and urine following a single smoked dose of cannabis. (2) Characterize the sensitivity, specificity, accuracy and length of detection of cannabinoids with the Draeger DrugTest 5000 after a single smoked dosed of cannabis. (3) Determine inter-matrix cannabinoid ratios in authentic specimens following controlled smoked cannabis. (4) Correlate cannabinoid concentrations in whole blood, plasma, breath, and oral fluid with impairment as determined through subjective assessments and neurocognitive tasks. (5) Determine stability over time of free and conjugated cannabinoids in urine from cannabis users following a single smoked dose of cannabis under various storage conditions.

Subject Population: Up to 50 healthy cannabis users aged 18-45 will be recruited for the study. In Part A, 10 completers with an average frequency of use of at least twice per month in the three months prior to study are required. In Part B, 10 occasional cannabis smokers with an average frequency of less than twice per week in the past three months and 10 chronic frequent cannabis smokers with an average frequency at least four times per week in the past three months are required.

Experimental Design and Methods: In parts A and B, participants smoke one standardized NIDA THC cigarette during a single visit. Serial blood and oral fluid collections (part A and B) and breath collections (part B only), and assessment of neurocognitive, physiological and subjective effects are performed once prior to and multiple times after smoking.

Outcome Measures: Primary outcome measures for part A include cannabinoid concentrations in whole blood, plasma, and oral fluid, stability of these concentrations over time, performance on neurocognitive tasks, and subjective assessments. Primary outcome measures for part B include cannabinoid concentrations in whole blood, plasma, breath, and oral fluid, evaluation of the DrugTest 5000 and correlation of cannabinoid breath concentration with performance on neurocognitive tasks and subjective assessments. An outcome measure for subsequent occasional smoker participants after the 9th completer is stability over time of cannabinoid concentrations in whole blood and plasma collected in gray-top Vacutainer tubes containing sodium fluoride and potassium oxalate.

Benefits: There is no direct benefit to participants, but the study is likely to yield generalizable knowledge regarding cannabinoid pharmacokinetics, and pharmacodynamics for both Part A and Part B.

Risks: Participation in this study represents more than minimal risk for both Part A and Part B because of the administration of smoked cannabis.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 18 to 45 years of age;
  2. Cannabis use with a minimum frequency of at least twice per month during the three months prior to study entry for Part A or average frequency of cannabis smoking of less than twice per week (occasional cannabis smoker) in the past 3 months or at least four times per week (chronic frequent cannabis smoker) in the past 3 months for Part B;
  3. A positive urine cannabinoid screen if in the chronic frequent cannabis smoker group;
  4. Peripheral veins suitable for repeated venipuncture and/or placement of an intravenous catheter;
  5. Blood pressure (BP) and heart rate (HR) at or below the following values while sitting after five min rest: Systolic BP (SBP) 140 mm Hg, diastolic BP (DBP) 90 mm Hg, heart rate (HR) 100 bpm;
  6. ECG and three-minute rhythm strip without clinically relevant abnormalities;

EXCLUSION CRITERIA:

1. History or presence of any clinically significant illness, as detected by history, physical examination, and/or laboratory tests, that might put the subject at increased risk of adverse events;
2. History of a clinically significant adverse event associated with cannabis intoxication;
3. Donation of more than 450 mL of blood within 30 days of study drug administration;
4. If female, pregnant or nursing;
5. Currently interested in or participating in drug abuse treatment, or participated in drug abuse treatment within 60 days preceding study enrollment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2010-01-22; Study Completion 2013-11-29 (Actual)

PRIMARY OUTCOMES:
THC and metabolite concentrations in whole blood, plasma, and oral fluid, stability of these concentrations over time, performance on neurocognitive tasks and subjective assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Huestis, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

REFERENCES:
- [Background] Vega WA, Aguilar-Gaxiola S, Andrade L, Bijl R, Borges G, Caraveo-Anduaga JJ, DeWit DJ, Heeringa SG, Kessler RC, Kolody B, Merikangas KR, Molnar BE, Walters EE, Warner LA, Wittchen HU. Prevalence and age of onset for drug use in seven international sites: results from the international consortium of psychiatric epidemiology. Drug Alcohol Depend. 2002 Dec 1;68(3):285-97. doi: 10.1016/s0376-8716(02)00224-7. PMID 12393223
- [Background] Huestis MA, Gorelick DA, Heishman SJ, Preston KL, Nelson RA, Moolchan ET, Frank RA. Blockade of effects of smoked marijuana by the CB1-selective cannabinoid receptor antagonist SR141716. Arch Gen Psychiatry. 2001 Apr;58(4):322-8. doi: 10.1001/archpsyc.58.4.322. PMID 11296091
- [Background] Huestis MA. Pharmacokinetics and metabolism of the plant cannabinoids, delta9-tetrahydrocannabinol, cannabidiol and cannabinol. Handb Exp Pharmacol. 2005;(168):657-90. doi: 10.1007/3-540-26573-2_23. PMID 16596792